CLINICAL TRIAL: NCT07378696
Title: Implementing Evidence-Based Nursing: Leadership and Organizational Change for Implementation
Acronym: LOCI-FIN-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaakko Varpula (Other)
Responsible Party: Sponsor-Investigator, Jaakko Varpula, Postdoctoral researcher, University of Turku
Organization: University of Turku (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TY/1603/2025
Record Dates: First submitted 2026-01-14; First posted 2026-01-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Leadership; Self-Harm; Malnutrition Elderly
Keywords: Implementation; Evidence-based practice; Nursing; Leadership
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Leadership; Organizational Innovation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leadership and Organizational Change for Implementation (LOCI) (Experimental): LOCI (Leadership and Organizational Change for Implementation) is a structured leadership and organizational development strategy designed to help managers strengthen their skills in implementing evidence-based practices. It combines leadership training, individualized mentoring, and organizational support to create a workplace climate that makes it easier to adopt and sustain new, research-based ways of working.
  Interventions: Behavioral: Leadership and organizational change for implementation

INTERVENTIONS:
Behavioral: Leadership and organizational change for implementation — LOCI (Leadership and Organizational Change for Implementation) is a structured leadership and organizational development strategy designed to help managers strengthen their skills in implementing evidence-based practices. It combines leadership training, individualized mentoring, and organizational support to create a workplace climate that makes it easier to adopt and sustain new, research-based ways of working.

SUMMARY:
This study aims to find out whether a leadership and organizational development program called the LOCI (Leadership and Organizational Change for Implementation) strategy can help nurses and their managers use the best available research in everyday care. Using evidence-based practice.

Previous work in the region showed that nurses and their managers want to use evidence-based practices but face challenges, such as unclear processes, limited support, and differences in skills. The LOCI strategy has helped leaders in other countries improve how new practices are introduced and supported. This study will test a version of LOCI adapted for Finnish healthcare settings.

Nurse managers and staff from selected hospital and elder care units will:

Take part in leadership and training sessions. Receive individual and group mentoring. Work with their teams on plans that support introducing new, research-based ways of working.

Two evidence-based practices will be introduced:

In psychiatric units: A safety planning method to help prevent suicide among people receiving mental health care.

In elder care units: Better ways to identify and treat malnutrition among older adults.

The study involves:

Nurse managers Nursing staff Senior nurse leaders Specialist nurses who support the training

The study will run for one year. The LOCI program lasts nine months, followed by a three-month follow-up period.

Assessment:

How well the adapted LOCI strategy works in practice (for example, whether participants find it useful).

Whether leadership skills and workplace support for evidence-based practices improve.

Whether the new care practices (suicide safety planning and malnutrition prevention) are used more often and more effectively.

Participants will complete questionnaires, take part in interviews or group discussions, and researchers will review documentation and care records to understand how the changes progress.

The study may help improve leadership skills, strengthen support for evidence-based practice, and improve care for patients in both mental health and elder care settings. The results may also help other healthcare organizations adopt similar approaches.

The study follows strict ethical and data protection rules. Survey participation is voluntary, and all personal information will be handled securely and confidentially. The care practices being introduced are already recommended in Finland and are part of normal care.

ELIGIBILITY:
Inclusion Criteria:

* Nurse manager
* Registered nurse
* Practical nurse
* Nurse director

Exclusion Criteria:

• Other healtcare professionals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 3months after start of intervention, 9 months (end of intervention)
  Acceptability of Intervention Measure (AIM), 4-item, 5-point Likert Scale (1-5), Min score 5, Max score 20. Higher scores indicate greater acceptability.
Appropriateness | 3months after start of intervention, 9 months (end of intervention)
  Intervention Appropriateness Measure (IAM), 4-item, 5-point Likert scale (1-5), Min score 5, Max score 20. Higher scores indicate greater appropriateness.
Feasibility of intervention | 3months after start of intervention, 9 months (end of intervention)
  Feasibility of Intervention Measure (FIM), 4-item, 5-point Likert scale (1-5), Min score 5, Xax score 20. Higher scores indicate greater feasibility.

SECONDARY OUTCOMES:
Effectiveness to implementation leadership | Baseline, 3month, 8months, 3 month follow-up
  Implementation leadership scale (ILS), 21-item, 5-point Likert scale (0-4). Min 0 and Max score 84. Higher scores indicate better implementation-supportive leadership.
Effectiveness to transformational leadership | Baseline, 3month, 8months, 3 month follow-up
  Global Transformational Leadership Scale (GTL), 7-item, 5-point Likert Scale (1-5), Min 7, Max score 35, higher score indicate better outcome, more transformational leadership behaviours.
Effectiveness to implementation climate | Baseline, 3month, 8months, 3 month follow-up
  Implementation Climate Scale (ICS), 27-item, 5-point Likert scale (0-4), Min 0, Max score 108, higher scores indicate better outcomes - stronger organizational climate supporting evidence-based practice implementation.
Effectiveness to evidence-based practice attitudes | Baseline, 3month, 8months, 3 month follow-up
  The Evidence-based Practice Attitude Scale (EBPAS), 15-item, 5-point Likert Scale (0-4). Min 0, Max score 60, higher scores indicate better outcome, more positive atittudes towards evidence-based practice.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Axelin, Professor, Study Director — University of Turku, Department of Nursing Science
Locations (1):
- The Wellbeing Services Country of Southwest Finland, Turku, Finland

IPD SHARING:
Plan to Share IPD: Yes
De-identified instrument-level data derived from questionnaires (ILS, GTL, ICS, EBPAS, AIM, IAM, FIM) completed by staff participants will be shared. These datasets will include item-level responses but will exclude any direct identifiers or variables that could reasonably enable re-identification.
Time Frame: Instrument-level IPD will be made available upon publication of the main study findings.
Access Criteria: Researchers may request access by contacting the principal investigators. Data will be shared through a secure repository after approval of a brief data-use proposal and signing a data-use agreement.